CLINICAL TRIAL: NCT02295462
Title: Effect of Person-Centred-Care on Antipsychotic Drug Use in Nursing Homes: a Cluster-randomised Trial
Acronym: EPCentCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: University of Luebeck (Other); University of Witten/Herdecke (Other)
Responsible Party: Principal Investigator, Gabriele Meyer, Prof. Dr., Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EPCentCare; 01GY1335A (Other Grant/Funding Number: German Federal Ministry of Education and Research); 01GY1335B (Other Grant/Funding Number: German Federal Ministry of Education and Research); 01GY1335C (Other Grant/Funding Number: German Federal Ministry of Education and Research)
Record Dates: First submitted 2014-11-12; First posted 2014-11-20 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Dementia
Keywords: nursing homes; person-centered care; inappropriate prescriptions; cluster-randomised controlled trial; antipsychotic drugs
MeSH Terms: conditions — Dementia | interventions — Patient-Centered Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Person-centered Care (Experimental): Medication Review + Person-centered Care
  Interventions: Other: Person-centered Care; Other: Optimised Treatment
- Optimised Treatment (Active Comparator): Medication Review
  Interventions: Other: Optimised Treatment

INTERVENTIONS:
Other: Person-centered Care — Medication Review + Person-centered Care
  Arms: Person-centered Care
Other: Optimised Treatment — Medication Review only

SUMMARY:
Background: Up to 90% of nursing home residents with dementia experience behavioural and psychological symptoms like apathy, agitation, and anxiety. According to analyses of prescription prevalence in Germany, antipsychotic drugs seem to be prescribed as first line treatment of neuropsychiatric symptoms in persons with dementia. A huge number is prescribed for inappropriate reasons and too long without regular review. The use of antipsychotics is associated with adverse events like increased risk of falling, stroke, and mortality. This study aims to investigate whether a person-centered care approach developed in the United Kingdom can be adapted and implemented in German nursing homes. The aim of the investigators trial is to achieve a clinically relevant reduction of the proportion of residents with alt least one antipsychotic drug prescription.

Methods/Design: Cluster-randomised controlled trial comparing an intervention group (two-day initial skill training on person-centred care and on-going training and support programme) with a control group receiving optimised usual care. Both study groups will receive a medication review by an experienced psychiatrist with feedback to the prescribing physician. Overall, 36 nursing homes from East, North and West Germany will be included and randomised. The primary outcome is defined as the proportion of residents receiving at least one antipsychotic medication at 12 months. Secondary outcomes are residents' quality of life, behavioural and psychological symptoms of dementia as well as safety parameters like falls and fall-related medical attention. Cost parameters will be collected and process evaluation will be performed alongside the trial.

ELIGIBILITY:
On cluster level

Inclusion Criteria:

* nursing homes with at least 50 residents

Exclusion Criteria:

* other ongoing trial in the institution

On individual level

Inclusion Criteria:

* all residents within a cluster are eligible to participate in the study

Exclusion Criteria:

* diagnoses of schizophrenia, schizoaffective psychosis, or other forms of primary psychosis
* respite care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1158 (Actual)
Dates: Start 2014-12; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Proportion of residents receiving at least one antipsychotic medication after 12 months | 12 months

SECONDARY OUTCOMES:
Residents' quality of life | 12 months
  Will be measured with the QoL-AD
Behavioural and psychological symptoms of dementia | 12 months
  Will be measured with the CMAI
Costs within trial period | 12 months
  Cost parameters will be collected alongside the trial on intervention-related components as well as outcome-related components. Costs which are explicitly trial-associated will not be taken into account for cost analysis.
Falls and fall-related medical attention | 12 months
Physical restraints within study period | 12 months
  Physical restraints will be assessed retrospectively by data extraction from residents' records- The following devices will be assessed: bilateral bedrails, belts, fixed tables, and other measures limiting free body movement.
Median daily dose of antipsychotics in chlorpromazine equivalents within study period | 12 months
  Each resident's daily dose of antipsychotic drugs will be translated into chlorpromazine daily equivalents.

OTHER OUTCOMES:
Process evaluation | 12 months
  Different methods will be used for data collection: investigators documentation, questionnaires on staff knowledge and self-efficacy, structured interviews and in depth-interviews with staff.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Meyer, Prof. Dr., Principal Investigator — Martin-Luther-Universität Halle-Wittenberg
Locations (3):
- Germany (3):
  - Universität Witten/Herdecke, Witten Herdecke, North Rhine-Westphalia
  - Martin-Luther-Universität Halle-Wittenberg, Halle, Saxony-Anhalt
  - University of Luebeck, Lübeck, Schleswig-Holstein

REFERENCES:
- [Derived] Richter C, Fleischer S, Langner H, Meyer G, Balzer K, Kopke S, Sonnichsen A, Loscher S, Berg A. Factors influencing the implementation of person-centred care in nursing homes by practice development champions: a qualitative process evaluation of a cluster-randomised controlled trial (EPCentCare) using Normalization Process Theory. BMC Nurs. 2022 Jul 8;21(1):182. doi: 10.1186/s12912-022-00963-6. PMID 35804407
- [Derived] Richter C, Berg A, Langner H, Meyer G, Kopke S, Balzer K, Wolschon EM, Silies K, Sonnichsen A, Loscher S, Haastert B, Icks A, Wolf U, Fleischer S. Effect of person-centred care on antipsychotic drug use in nursing homes (EPCentCare): a cluster-randomised controlled trial. Age Ageing. 2019 May 1;48(3):419-425. doi: 10.1093/ageing/afz016. PMID 30806453
- [Derived] Dichter MN, Wolschon EM, Schwab CGG, Meyer G, Kopke S. Item distribution and inter-rater reliability of the German version of the quality of life in Alzheimer's disease scale (QoL-AD) proxy for people with dementia living in nursing homes. BMC Geriatr. 2018 Jun 19;18(1):145. doi: 10.1186/s12877-018-0834-z. PMID 29914389
- [Derived] Richter C, Berg A, Fleischer S, Kopke S, Balzer K, Fick EM, Sonnichsen A, Loscher S, Vollmar HC, Haastert B, Icks A, Dintsios CM, Mann E, Wolf U, Meyer G. Effect of person-centred care on antipsychotic drug use in nursing homes (EPCentCare): study protocol for a cluster-randomised controlled trial. Implement Sci. 2015 Jun 4;10:82. doi: 10.1186/s13012-015-0268-3. PMID 26037324